CLINICAL TRIAL: NCT06018207
Title: The Median Effective Dose of Midazolam Oral Solution for Preoperative Hypnosis in Non-Elderly Adults in the Preoperative Room: An Up-and-Down Sequential Allocation Trial
Brief Title: ED50 of Midazolam Oral Solution for Preoperative Hypnosis in Adults : An Up-and-Down Sequential Allocation Trial
Acronym: ED50-MOS-PH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZSLYEC-402
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Dose; Midazolam; Preoperative
Keywords: midazolam; sleep; ED50; ED95; preoperative room;adult
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- An Up-and-Down Sequential Allocation (Experimental): An Up-and-Down Sequential Allocation is that the dose is varied based on the hypnosis response of the previous patient after taking midazolam oral solution for 1 hour.
  Interventions: Drug: Midazolam oral solution

INTERVENTIONS:
Drug: Midazolam oral solution — The ED50 dose of midazolam oral solution for hypnosis is studied using an up-and-down sequential allocation while waiting for surgery and general anesthesia in preoperative room.
  The starting dose is 6 mg and the step size is 1 mg. The interval sequential dose is varied by 1 mg based on the hypnosis response of the previous patient after one hour.
  Definition of successful hypnosis by taking midazolam oral solution:
  The polysomnograph (PSG) not only shows stage N2 within 30 minutes, but also shows stage N3 within an hour; or else, definition of unsuccessful hypnosis.
  The procedure is as follows: (1) The first subject is given 6mg of midazolam oral solution; (2) If succeed, the second subject takes 5mg; (3) If not succeed, the second subject takes 7mg; (4) Until seven sequence reversal inflection points.

SUMMARY:
Due to sleep deficiency, patients with insomnia syndrome or sub-clinical insomnia syndrome often undergo severe stress while waiting for surgery. Studies have reported that preoperative hypnosis could reduce stress and promote recovery. Midazolam has been recommended to patients who under severe stress for preoperative sedation and anti-anxiety. However, midazolam for preoperative hypnosis monitored with polysomnography (PSG) has not been studied. In this exploratory study, the median effective dose (ED50) and ED95 of Midazolam Oral Solution for preoperative hypnosis in non-elderly adults using the gold standard tool of PSG, will be explored by up-and-down sequential allocation and probit method.

DETAILED DESCRIPTION:
The exploratory study of ED50 will be manipulated by an up-and-down sequential allocation with a single arm prospectively.

1. The day before surgery, subjects will be enrolled according to the inclusion criteria and sign the informed consent voluntarily.
2. On the day of surgery, the clinical process is as follows. According to the routine medical procedures of our center, patients should access in the operating room about 2 hours before their surgery for adequate preparation.After peripheral venous catheterization, monitored by electrocardiogram, noninvasive blood pressure, and pulse oxygen saturation, invasive procedures,such as arterial catheterization, central venous catheterization or nerve blocks, will be operated individually according to surgical and anesthesia necessity.
3. The intervention of Midazolam Oral Solution for preoperative hypnosis will be done after invasive procedures. The ED50 dose of midazolam oral solution for hypnosis is studied using an up-and-down sequential allocation while waiting for surgery and general anesthesia in preoperative room.

   The starting dose is 6 mg and the step size is 1 mg. The interval sequential dose is varied by 1 mg based on the hypnosis response of the previous patient after one hour. Sleep of the subjects will be monitored by portable PSG (Alice PDx).

   Definition of successful hypnosis by taking midazolam oral solution: The polysomnograph (PSG) not only shows stage N2 within 30 minutes, but also shows stage N3 within an hour; or else, definition of unsuccessful hypnosis. The intervention procedure : (1) The first subject takes 6mg of midazolam oral solution; (2) If succeed, the second subject will take 5mg; (3) If not succeed, the second subject will take 7mg; (4) Until seven sequence reversal inflection points.
4. Measures of safety assurance:

(1)Monitoring: Electrocardiogram, blood pressure, pulse oxygen saturation, respiratory rate, consciousness; (2)Monitors, negative pressure suction devices, oxygen inhalation devices, ventilators, items needed for emergency airway establishment, first aid medications, systemically trained anesthesiologists and nurses; (3)Emergencies include, but are not limited to: vomiting, respiratory depression, and respiratory obstruction. If any of the above events occur after intervention, the clinical procedures or emergency procedures will be followed immediately.

Statistics： Using the sequential and probit method to determine the median effective dose and ED95. The sample size is considered adequate once 7 pairs of sequence reversals have been reached. Based on the preliminary test analysis, it is anticipated that 40 subjects would be required.

ELIGIBILITY:
Inclusion Criteria:

1. Signed of informed consent voluntarily;
2. Native Chinese speaker;
3. Age 18-60 years old, male or female;
4. BMI 18-30 kg/m2;
5. American Society of Anesthesiologists (ASA) grade 1 or 2, New York Heart Association (NYHA) gradeⅠorⅡ;
6. Non-emergency cancer resection surgery is planned in the next day;
7. Insomnia syndrome or sub-clinical insomnia syndrome in the past 1 month.

Exclusion Criteria:

1. Contraindications for Midazolam Oral Solution (According to the Instruction for Midazolam Oral Solution);
2. High risk of Obstructive Sleep Apnea Symptoms (Total score of STOP-Bang scale ≥3 points);
3. Suspected dementia (Total score of Mini-Mental State Examination (MMSE) according to years of education: 0 year≤19 points; 1~6 years≤22 points; above of 6 years≤26 points);
4. Severe depressive symptom within two weeks (Total score of Patient Health Questionnaire-9 (PHQ-9)≥15);
5. History of Neurological and Psychiatric diseases (According to the electronic medical record system);
6. History of Chronic Obstructive Pulmonary Disease (According to the electronic medical record system);
7. History of Heart Failure (According to the electronic medical record system);
8. Intestinal obstruction(The electronic medical record system records those who currently have any type of intestinal obstruction);
9. Liver and renal insufficiency;
10. Have taken opioids or drugs that act on the central nervous system within one week;
11. Take CYP3A4 isoenzyme inhibitors or inducers within one week (According to the Instruction for Midazolam Oral Solution);
12. Consume any alcoholic beverage within 24 hours;
13. Substance abusers (including alcohol, drugs or addictive substances);
14. Pregnant or lactating women;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
The Median Effective Dose (ED50) of Midazolam Oral Solution | Within 1 hour after taking Midazolam Oral Solution while waiting for surgery in the operating room
  The Median Effective Dose (ED50) of Midazolam Oral Solution for Preoperative Hypnosis in Non-Elderly Adults in the Preoperative Room, using an up-and-down sequential allocation.

SECONDARY OUTCOMES:
ED95 of Midazolam Oral Solution for Preoperative Hypnosis in Non-Elderly Adults in the Preoperative Room | Within 1 hour after taking Midazolam Oral Solution while waiting for surgery in the operating room
  ED95 of Midazolam Oral Solution for Preoperative Hypnosis in Non-Elderly Adults in the Preoperative Room, using an up-and-down sequential allocation and calculating by Probit method (probability unit regression).
Description of Proportions of stage N1 in different doses | Within 1.5 hour after taking Midazolam Oral Solution while waiting for surgery in the operating room
  We speculate that the sleep structure is different with the different doses of Midazolam Oral Solution.
  Description of Proportions of stage N1 in different doses. Data are expressed as percentages.
Description of Proportions of stage N2 in different doses | Within 1.5 hour after taking Midazolam Oral Solution while waiting for surgery in the operating room
  We speculate that the sleep structure is different with the different doses of Midazolam Oral Solution.
  Description of Proportions of stage N2 in different doses. Data are expressed as percentages.
Description of Proportions of stage N3 in different doses | Within 1.5 hour after taking Midazolam Oral Solution while waiting for surgery in the operating room
  We speculate that the sleep structure is different with the different doses of Midazolam Oral Solution.
  Description of Proportions of stage N3 in different doses. Data are expressed as percentages.
Description of Proportions of stage REM in different doses | Within 1.5 hour after taking Midazolam Oral Solution while waiting for surgery in the operating room
  We speculate that the sleep structure is different with the different doses of Midazolam Oral Solution.
  Description of Proportions of stage REM in different doses. Data are expressed as percentages.
Description of Sleep latency(min) in different doses | Within 1 hour after taking Midazolam Oral Solution while waiting for surgery in the operating room
  Sleep latency(min): the time it takes from taking Midazolam Oral Solution to entering the N2 phase of sleep.
  We speculate that sleep latency is different with the doses of Midazolam Oral Sulution.
  Data are expressed as mean ± standard deviation.
Description of anti-anxiety effects in different doses | Within 1.5 hour after taking Midazolam Oral Solution while waiting for surgery in the operating room
  Description of the different anti-anxiety effects between those who reach the hypnotic end point and those who do not, using the Generalized Anxiety Disorder-2 (GAD-2) scale.
  Data are expressed as mean ± standard deviation.
Description of sedative effect in different doses | Within 1.5 hour after taking Midazolam Oral Solution while waiting for surgery in the operating room
  Description of the different sedative effects between those who reach the hypnotic end point and those who do not, using Richmond Agitation and Sedation Scale (RASS).
  Data are expressed as mean ± standard deviation.
Description of satisfaction for preoperative hypnosis in different doses | On postoperative day 1
  Description of sleep satisfaction while waiting for surgery in the operating room after taking Midazolam Oral Solution, using Visual Analogue Scale（VAS）score (0-10 points).
  Data are expressed as mean ± standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Jin sanqing, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No